CLINICAL TRIAL: NCT02912286
Title: Postoperative Pain Following Irrigation With Endodontic Needle, Sonic and Passive Ultrasonic Techniques: A Randomized Controlled Trial
Brief Title: Postoperative Pain Following Irrigation With Endodontic Needle, Sonic and Passive Ultrasonic Techniques
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nancy Samy, Assisstant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEBD-CU-2016-09-200
Record Dates: First submitted 2016-09-20; First posted 2016-09-23 (Estimated); Last update posted 2016-09-23 (Estimated); Status verified 2016-09

CONDITIONS: Tooth,Non-vital

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- conventional needle irrigation (Active Comparator): side-vented needle used for endodontic irrigation
  Interventions: Device: conventional needle irrigation
- passive ultrasonic irrigation (Experimental): IrriSafe ultrasonic tip used for irrigation agitation in endodontic treatment
  Interventions: Device: passive ultrasonic irrigation
- sonic irrigation (Experimental): Vibringe is a sonic irrigation system used to irrigate and activate the irrigant at same time
  Interventions: Device: sonic irrigation

INTERVENTIONS:
Device: conventional needle irrigation — conventional side-vented syringe used to deliver irrigant in root canal treatment
  Arms: conventional needle irrigation
Device: passive ultrasonic irrigation — ultrasonic tip (IrriSafe) activate the irrigant after mechanical preparation in root canal treatment
  Arms: passive ultrasonic irrigation
Device: sonic irrigation — vibringe system is a sonic device that deliver and agitate the irrigant
  Arms: sonic irrigation

SUMMARY:
The aim of this study is to compare the postoperative pain after root canal treatment following irrigation by endodontic needle, sonic and passive ultrasonic irrigation techniques.

DETAILED DESCRIPTION:
Different irrigation delivery systems are introduced to the market aiming to improve root canals disinfection. The conventional endodontic needle is commonly used because of its ease in use and good control of needle depth and irrigant volume. However it carries a higher risk of extruding the solution periapically because of positive pressure used in solution delivery.

Passive ultrasonic irrigation is a noncutting irrigation technique that is done with ultrasonically activated files with continuous or intermittent flow of irrigant. It was shown that it is effective in removing remnants of pulp tissue, dentin debris and planktonic bacteria.

The vibringe (Cavex Holland BV, Haarlem, the Netherlands) is an irrigation device that combines manual delivery and sonic activation of the irrigant.

The aim of this study is to compare the postoperative pain after root canal treatment following irrigation by endodontic needle, sonic and passive ultrasonic irrigation techniques.

ELIGIBILITY:
Inclusion Criteria:

* Males or Females
* Age between 16-60 years old
* Permanent Mandibular molars with:

  * Non-vital response of pulp tissue
  * Absence of spontaneous pain

Exclusion Criteria:

* Pregnant females
* Patients having significant systemic disorder
* Patients received analgesics, anti-inflammatory or antibiotic in the last 24 hours
* Teeth that have:

  * Vital pulp tissues
  * Association with swelling or fistulous tract
  * Acute periapical abscess
  * Greater than grade I mobility
  * Pocket depth greater than 5mm
  * Previous endodontic treatment

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 57 (Estimated)
Dates: Start 2017-01; Primary Completion 2019-01 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
postoperative pain measured by numerical rate scale | 4 hours after treatment
  Numerical rate scale (NRS) consists of a line graded from 0-10 where 0 indicates no pain and 10 indicates worst pain, patient will choose the number that describe his pain level.

IPD SHARING:
Plan to Share IPD: No